CLINICAL TRIAL: NCT05699590
Title: Galectin-3 Immunoreactivity in Papillary Thyroid Carcinoma
Brief Title: Galectin-3 in Papillary Thyroid Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amira Ahmed Abdelnaby, Lecturer of pathology, Sohag University
Other Study IDs: Soh-Med-23-1-35
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Galactin 3-thyroid Carcinoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Thyroid cancer is a common head and neck malignancy. It is the most common endocrine tumor in the body accounting for 1% of all cancers worldwide. The incidence of thyroid cancer varies worldwide. Most countries have reported an upward trend in its incidence.

Thyroid cancer encompass the most common well-differentiated papillary carcinoma (80% of all thyroid cancers) and follicular carcinoma (15%), as well as poorly differentiated carcinoma (< 1%) and anaplastic carcinoma (< 2%).

Papillary thyroid carcinomas (PTCs) are the most commonly encountered thyroid malignancies. The diagnosis of PTC is based on the special nuclear features such as overlapping of nuclei, intranuclear inclusions, optical clearing, anisonucleosis and nuclear grooves. However, it is often difficult to differentiate PTC from benign papillary thyroid hyperplasia . As differentiation between benign or malignant thyroid lesions has clinical, therapeutic, and prognostic significance, it is necessary to make accurate diagnosis by using biomarkers.

Recently, a large number of immunohistochemical (IHC) markers have been studied to assist in differentiating non-neoplastic lesions from malignant thyroid lesions. CK19, galectin-3, TG, Ki67, BRAF, calcitonin, HBME-1, TTF-1, and RET are some of the examples of these IHC markers.

Galectin-3 is a 31-kDa β-galactoside binding lectin. It has been shown to be expressed by several types of non-neoplastic and neoplastic cells, and it is involved in cell-cell adhesion and in cell-matrix interactions.

ELIGIBILITY:
Inclusion Criteria:

1. Thyroidectomy specimens both hemithyroidectomy and total thyroidectomy.
2. All the studied cases include sufficient materials for the immunohistochemical study.
3. Complete clinical data

Exclusion Criteria:

1. Patients with recurrence of the primary tumor.
2. Patients with a history of preoperative chemotherapy and/or radiotherapy.
3. Insufficient or tiny tissue biopsies

Ages: 20 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Formalin fixed and paraffin embedded prostatic tissue blocks from 70 patients
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Diagnosis and prognosis of papillary thyroid carcinoma both classic variant and follicular variant | Two or three days after staining tissue sections with Galactin 3 antibody
  evaluation of Galectin-3 Immunostaining in Papillary Thyroid Carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Amira Ahmed Abdelnaby, Lecturer, Principal Investigator — Pathology department, Faculty of medicine ,Sohag university

IPD SHARING:
Plan to Share IPD: Undecided